CLINICAL TRIAL: NCT06804265
Title: Molecular Biology (Multiplex PCR) in the Identification of Pathogens at Reimplantation in the Two-Stage Treatment of Periprosthetic Infections (PJI)
Brief Title: Molecular Biology in the Identification of Pathogens at Reimplantation in the Two-Stage Treatment of Periprosthetic Infections
Acronym: MOLPJI
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: MOLPJI
Record Dates: First submitted 2025-01-10; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-12

CONDITIONS: Periprosthetic Joint Infection (PJI)
Keywords: Multiplex PCR

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to measure the diagnostic accuracy of the Multiplex PCR technique in identifying pathogens during the diagnostic stage of resolving pre-implantation infection, in the context of treatment according to two-stage protocol for PJIs. This evaluation will be conducted by comparing the results obtained by Multiplex PCR with those derived from standard culture examination.

DETAILED DESCRIPTION:
The data that will be collected are:

1. Pre-implantation data: timing of infection, bacterial population involved, type of surgery (primary or revision implantation). Baseline characteristics of patients, such as gender, age, history of previous interventions (including date, number and type of interventions), comorbidities, ASA score, and lifestyle habits (such as smoking and alcohol) will also be recorded. Local problems of the operated limb and investigations performed, including instrumental and laboratory tests, will be documented.
2. Data on explant surgery and postoperative course: details of whether or not spacer cement was used according to the two-stage protocol, the type of spacer cement used, the occurrence of intraoperative complications and the characteristics and duration of postoperative antibiotic therapy will be recorded. Results of molecular investigations will be documented, both pre-operative on ultrasound aspirate, intraoperative and 15 days after discontinuation of antibiotic therapy. Results of histological and culture examinations of the preoperative and intraoperative aspirate, postoperative complications will be included.
3. Data related to reimplantation: timing of reimplantation, result of molecular, culture, and histological examinations on intraoperative specimens, post-reimplantation antibiotic therapy, intraoperative and postoperative complications, clinical status at follow-up (recurrence/persistence of infection), and duration of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of periprosthetic infection of hip, knee, shoulder on primary or already revised implant.
* treatment of infection with two-stage protocol.
* Obtaining informed consent
* Age ≥18 years

Exclusion Criteria:

* Isolates obtained during explantation not included in MULTIPLEX PCR panel

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The analysis will be performed on patients treated at the Department of Orthopaedics and Traumatology of IRCCS Azienda Ospedaliero Universitaria di Bologna, Policlinico di S.Orsola, from study approval until two years after study approval. The study population will be hip, knee and shoulder joint replacement patients diagnosed with PJI and undergoing prosthetic explantation surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-07 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Accuracy, sensitivity and specificity of the PCR technique in identifying the pathogen responsible for PJIs | up to 100 weeks
  comparison with the current diagnostic gold standard, represented by culture examination

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano - De Paolis, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy